CLINICAL TRIAL: NCT01098539
Title: A Randomized, Double-Blind, Active-Controlled, Parallel-Group, Multicenter Study to Determine the Efficacy and Safety of Albiglutide as Compared With Sitagliptin in Subjects With Type 2 Diabetes Mellitus With Renal Impairment
Brief Title: A Study of the Efficacy and Safety of Albiglutide in Subjects With Type 2 Diabetes With Renal Impairment.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 114130
Record Dates: First submitted 2010-04-01; First posted 2010-04-02 (Estimated); Results first posted 2014-05-16 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: sitagliptin; albiglutide; renal impairment
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency | interventions — rGLP-1 protein; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- albiglutide (Active Comparator): albiglutide weekly subcutaneous injection + sitagliptin matching placebo
  Interventions: Biological: albiglutide
- sitagliptin (Active Comparator): albiglutide matching placebo + sitagliptin
  Interventions: Drug: sitagliptin

INTERVENTIONS:
Biological: albiglutide — albiglutide weekly subcutaneous injection + sitagliptin matching placebo
  Arms: albiglutide
Drug: sitagliptin — albiglutide matching placebo + sitagliptin (25mg, 50mg or 100mg depending on level of renal impairment)
  Arms: sitagliptin

SUMMARY:
This randomized, double-blind, active-controlled study evaluates the efficacy and safety of a weekly dose of albiglutide as compared with sitagliptin. Subjects who are renally impaired with a historical diagnosis of type 2 diabetes mellitus and whose glycemia is inadequately controlled on their current regimen of diet and exercise or their antidiabetic therapy of metformin, thiazolidinedione, sulfonylurea, or any combination of these oral antidiabetic medications will be recruited into the study.

DETAILED DESCRIPTION:
This randomized, double-blind, active-controlled, 2 parallel-group, multicenter study evaluates the efficacy and safety of a weekly subcutaneously injected dose of albiglutide as compared with sitagliptin. Subjects who are renally impaired with a historical diagnosis of type 2 diabetes mellitus and whose glycemia is inadequately controlled on their current regimen of diet and exercise or their antidiabetic therapy of metformin, thiazolidinedione, sulfonylurea, or any combination of these oral antidiabetic medications will be recruited into the study.

ELIGIBILITY:
Inclusion Criteria:

* Renally impaired with a historical diagnosis of type 2 diabetes mellitus and is experiencing inadequate glycemic control on their current regime of diet and exercise or their antidiabetic therapy of metformin, TZD, SU, or any combination of these oral antidiabetic medications
* BMI >/=20 kg/m2 and </=45 kg/m2
* Fasting C-peptide >/=0.8 ng/mL (>/=0.26 nmol/L)
* HbA1c between 7.0% and 10.0%, inclusive.

Exclusion Criteria:

* History of cancer
* History of treated diabetic gastroparesis
* Current biliary disease or history of pancreatitis
* History of significant gastrointestinal surgery
* Recent clinically significant cardiovascular and/or cerebrovascular disease
* History of human immunodeficiency virus infection
* Abnormal liver function or acute symptomatic infection with hepatitis B or hepatitis C
* Female subject is pregnant (confirmed by laboratory testing), lactating, or <6 weeks postpartum
* Known allergy to any GLP 1 analogue, sitagliptin, other study medications' excipients, excipients of albiglutide, or Baker's yeast
* Receipt of any investigational drug or sitagliptin within the 30 days or 5 half lives, whichever is longer, before Screening or a history of receipt of an investigational antidiabetic drug within the 3 months before randomization or receipt of albiglutide in previous studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 507 (Actual)
Dates: Start 2010-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (186):
- United States (100):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Gulf Shores, Alabama
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Toney, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Los Gatos, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Dimas, California
  - GSK Investigational Site, Tarzana, California
  - GSK Investigational Site, West Hills, California
  - GSK Investigational Site, Whittier, California
  - GSK Investigational Site, Doral, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Miami Beach, Florida
  - GSK Investigational Site, New Port Richey, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Winter Park, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Blue Ridge, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Roswell, Georgia
  - GSK Investigational Site, Stone Mountain, Georgia
  - GSK Investigational Site, Valparaiso, Indiana
  - GSK Investigational Site, Des Moines, Iowa
  - GSK Investigational Site, Mission, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Paducah, Kentucky
  - GSK Investigational Site, Alexandria, Louisiana
  - GSK Investigational Site, Bangor, Maine
  - GSK Investigational Site, Hyattsville, Maryland
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Dearborn, Michigan
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Flint, Michigan
  - GSK Investigational Site, Saint Clair Shores, Michigan
  - GSK Investigational Site, Taylor, Michigan
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, North Massapequa, New York
  - GSK Investigational Site, Staten Island, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Hurst, North Carolina
  - GSK Investigational Site, Shelby, North Carolina
  - GSK Investigational Site, Tabor City, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Gallipolis, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Altoona, Pennsylvania
  - GSK Investigational Site, Downington, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, North Myrtle Beach, South Carolina
  - GSK Investigational Site, Taylors, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Franklin, Tennessee
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Tullahoma, Tennessee
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Deer Park, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Grapevine, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Humble, Texas
  - GSK Investigational Site, Hurst, Texas
  - GSK Investigational Site, Irving, Texas
  - GSK Investigational Site, Midland, Texas
  - GSK Investigational Site, North Richland Hills, Texas
  - GSK Investigational Site, Pearland, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, Richardson, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Schertz, Texas
  - GSK Investigational Site, Sugarland, Texas
  - GSK Investigational Site, Tomball, Texas
  - GSK Investigational Site, Bountiful, Utah
  - GSK Investigational Site, South Burlington, Vermont
  - GSK Investigational Site, Burke, Virginia
  - GSK Investigational Site, Manassas, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Salem, Virginia
  - GSK Investigational Site, Tacoma, Washington
- Australia (12):
  - GSK Investigational Site, Garran, Australian Capital Territory
  - GSK Investigational Site, Camperdown, New South Wales
  - GSK Investigational Site, Auchenflower, Queensland
  - GSK Investigational Site, Caboolture, Queensland
  - GSK Investigational Site, Herston, Queensland
  - GSK Investigational Site, Kippa-Ring, Queensland
  - GSK Investigational Site, Box Hill, Victoria
  - GSK Investigational Site, Clayton, Victoria
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Parkville, Victoria
  - GSK Investigational Site, Fremantle, Western Australia
- Brazil (4):
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, São Paulo, São Paulo
  - GSK Investigational Site, Brasília
  - GSK Investigational Site, Mogi das Cruzes
- Colombia (3):
  - GSK Investigational Site, Barrangquilla
  - GSK Investigational Site, Bogotá
  - GSK Investigational Site, Floridablanca-Santander
- Germany (5):
  - GSK Investigational Site, Bad Nauheim, Hesse
  - GSK Investigational Site, Bad Lauterberg im Harz, Lower Saxony
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Berlin, State of Berlin
- India (8):
  - GSK Investigational Site, Ahmedabad
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Belagavi
  - GSK Investigational Site, Chennai
  - GSK Investigational Site, Lucknow
  - GSK Investigational Site, Manipal
  - GSK Investigational Site, Mumbai
  - GSK Investigational Site, Nashik
- Israel (6):
  - GSK Investigational Site, Ashkelon
  - GSK Investigational Site, Beersheba
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Holon
  - GSK Investigational Site, Kfar Saba
  - GSK Investigational Site, Safed
- Peru (7):
  - GSK Investigational Site, Arequipa, Arequipa
  - GSK Investigational Site, Ica, Ica
  - GSK Investigational Site, Lima, Lima Province
  - GSK Investigational Site, Callao, Lima
  - GSK Investigational Site, Piura, Piura
  - GSK Investigational Site, Lima
  - GSK Investigational Site, Trujillo
- Philippines (5):
  - GSK Investigational Site, Cebu City
  - GSK Investigational Site, Iloilo City
  - GSK Investigational Site, Makati City
  - GSK Investigational Site, Pasay
  - GSK Investigational Site, Tagbilaran City
- Russia (4):
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, St'Petersburg
  - GSK Investigational Site, Yaroslavl
- South Africa (10):
  - GSK Investigational Site, Port Elizabeth, Eastern Cape
  - GSK Investigational Site, Johannesburg, Gauteng
  - GSK Investigational Site, Lenasia, Gauteng
  - GSK Investigational Site, Pretoria, Gauteng
  - GSK Investigational Site, Durban, KwaZulu-Natal
  - GSK Investigational Site, Phoenix, KwaZulu-Natal
  - GSK Investigational Site, Houghton Estate
  - GSK Investigational Site, Pretoria
  - GSK Investigational Site, Somerset West
  - GSK Investigational Site, Tygerberg
- South Korea (3):
  - GSK Investigational Site, Seongnam-si
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon, Kyonggi-do
- Spain (7):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Torrevieja (Alicante)
- Taiwan (3):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Tainan
- United Kingdom (9):
  - GSK Investigational Site, Coventry, West Midlands
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Hertfordshire
  - GSK Investigational Site, Hull
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, Livingston
  - GSK Investigational Site, London
  - GSK Investigational Site, Plymouth
  - GSK Investigational Site, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- [Derived] Young MA, Wald JA, Matthews JE, Scott R, Hodge RJ, Zhi H, Reinhardt RR. Clinical pharmacology of albiglutide, a GLP-1 receptor agonist. Postgrad Med. 2014 Nov;126(7):84-97. doi: 10.3810/pgm.2014.11.2836. PMID 25387217
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 114130 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114130 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114130 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114130 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114130 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114130 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114130 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants entered into 2 weeks of Pre-screening and Screening; 4 weeks of Run-in/stabilization; 52-week Treatment Period for evaluation of efficacy and safety and 8 weeks of post treatment Follow-up. A total of 771 participants were screened, 507 were randomized and 495 received at least one dose of study treatment.
Groups:
- Albiglutide 30 mg: Participants received albiglutide 30 milligrams (mg) once weekly subcutaneously from Baseline until Week 52, with optional up-titration to 50 mg if additional glycemic control was required. Albiglutide was injected subcutaneously into the abdomen, on alternating right and left sides of the body. Participants also received sitagliptin matching placebo once daily orally. Participants who qualified for hyperglycemia rescue, on or after Week 2, continued in the study after rescue and continued to receive study treatment until study completion.
- Sitagliptin 100 mg: Participants with normal renal function (estimated glomerular filtration rate [eGFR] >89 milliliters per minute [mL/min]) received a sitagliptin 100 mg overcoated tablet once daily orally from Baseline until Week 52. The dose of sitagliptin was adjusted in a range of 25-100 mg based on the participant's severity of renal impairment using the modification of diet in renal disease (MDRD) formula. Participants also received albiglutide matching placebo once weekly subcutaneously from Baseline until Week 52. Albiglutide matching placebo was injected subcutaneously into the abdomen, on alternating right and left sides of the body. Participants who qualified for hyperglycemia rescue, on or after Week 2, continued in the study after rescue and continued to receive study treatment until study completion.
Period: Overall Study
Arm/Group | Albiglutide 30 mg | Sitagliptin 100 mg
Started | 249 | 246
Completed | 198 | 178
Not Completed | 51 | 68
Not completed — Adverse Event | 26 | 26
Not completed — Protocol Violation | 1 | 4
Not completed — Noncompliance | 3 | 5
Not completed — Lost to Follow-up | 4 | 4
Not completed — Withdrawal by Subject | 12 | 26
Not completed — Physician Decision | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Albiglutide 30 mg | Sitagliptin 100 mg | Total
Number analyzed (Participants) | 249 | 246 | 495
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.2 (8.37) | 63.5 (9.02) | 63.3 (8.69)
Gender [Count of Participants; unit: Participants]
  Female | 113 | 116 | 229
  Male | 136 | 130 | 266
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 36 | 42 | 78
  American Indian or Alaskan Native | 16 | 16 | 32
  Asian - Central/South Asian Heritage | 45 | 33 | 78
  Asian - East Asian Heritage | 26 | 29 | 55
  Asian - South East Asian Heritage | 13 | 14 | 27
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White - Arabic/North African Heritage | 0 | 1 | 1
  White - White/Caucasian/European Heritage | 112 | 111 | 223

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 26
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over a 2- to 3-month period. The Baseline HbA1c value is defined as the last non-missing value before the start of treatment. Change from Baseline in HbA1c was calculated as the value at Week 26 minus the value at Baseline. The analysis was performed using an Analysis of Covariance (ANCOVA) model with treatment group, region, history of prior myocardial infarction (yes versus no), and age category (<65 years versus >=65 years) as factors and Baseline HbA1c as a continuous covariate. The last observation carried forward (LOCF) method was used to impute missing data, in which the last non-missing post-Baseline on-treatment measurement was used to impute the missing measurement. If a participant had missing observation(s) immediately after Baseline, the Baseline observation was not carried forward and was left as missing.
Time Frame: Baseline; Week 26
Population: Intent-to-Treat (ITT) Population: all participants who received at least one dose of study medication and who had at least one post-Baseline assessment of the primary endpoint, HbA1c. Only those participants available at the indicated time point were assessed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c in the blood
Arm/Group | Albiglutide 30 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 242 | 236
Percentage of HbA1c in the blood | -0.83 (0.062) | -0.52 (0.063)
Statistical Analysis 1: Comparison: Albiglutide 30 mg vs Sitagliptin 100 mg; Test type: Non-Inferiority or Equivalence — The p-value was from a 1-sided t test to test whether the difference of LS means (albiglutide - sitagliptin) was less than or equal to the prespecified noninferiority margin of 0.4%; p < 0.0001, t-test, 1 sided; Median Difference (Final Values) = -0.32, 95% CI 2-sided [-0.49 to -0.15]

2. Secondary Outcome: Mean Change From Baseline in HbA1c at Weeks 4, 8, 12, 16, and 20: LOCF
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over a 2- to 3-month period. The Baseline HbA1c value is defined as the last non-missing value before the start of treatment. Change from Baseline in HbA1c was calculated as the post-Baseline value minus the Baseline value. The LOCF method was used to impute missing data, in which the last non-missing post-Baseline on-treatment measurement was used to impute the missing measurement. If a participant had missing observation(s) immediately after Baseline, the Baseline observation was not carried forward and was left as missing. Participants were analyzed in a particular treatment week if they had received at least one dose in that treatment week.
Time Frame: Baseline; Weeks 4, 8, 12, 16, and 20
Population: ITT Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c in the blood
Arm/Group | Albiglutide 30 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 246 | 240
Percentage of HbA1c in the blood
  Week 4, n=237, 234 | -0.43 (0.460) | -0.37 (0.512)
  Week 8, n=242, 236 | -0.60 (0.663) | -0.52 (0.785)
  Week 12, n=242, 236 | -0.69 (0.840) | -0.56 (0.989)
  Week 16, n=242, 236 | -0.75 (0.886) | -0.56 (1.103)
  Week 20, n=242, 236 | -0.79 (0.890) | -0.54 (1.083)

3. Secondary Outcome: Mean Change From Baseline in HbA1c at Weeks 4, 8, 12, 16, 20, 26, 36, 48, and Week 52: Observed Cases
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over a 2- to 3-month period. The Baseline HbA1c value is defined as the last non-missing value before the start of treatment. Change from Baseline in HbA1c was calculated as the post-Baseline value minus the Baseline value. The Observed Cases (OC) method (no imputation of missing data) was used. If a participant had missing observation(s) immediately after Baseline, the Baseline observation was not carried forward and was left as missing. Participants were analyzed in a particular treatment week if they had received at least one dose in that treatment week.
Time Frame: Baseline; Weeks 4, 8, 12, 16, 20, 26, 36, 48, and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c in the blood
Arm/Group | Albiglutide 30 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 246 | 240
Percentage of HbA1c in the blood
  Week 4, n=233, 228 | -0.43 (0.463) | -0.37 (0.512)
  Week 8, n=222, 213 | -0.63 (0.677) | -0.56 (0.794)
  Week 12, n=224, 216 | -0.71 (0.832) | -0.62 (0.940)
  Week 16, n=218, 209 | -0.75 (0.885) | -0.63 (1.085)
  Week 20, n=207, 196 | -0.86 (0.852) | -0.71 (0.931)
  Week 26, n=202, 178 | -0.93 (0.806) | -0.80 (0.887)
  Week 36, n=192, 155 | -1.01 (0.808) | -0.82 (1.014)
  Week 48, n=172, 139 | -1.01 (0.884) | -0.89 (0.977)
  Week 52, n=157, 118 | -1.04 (0.796) | -1.03 (0.883)

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 26
Description: The FPG test measures blood sugar levels after the participant has not eaten (fasted) for 12 to 14 hours. The Baseline FPG value is define as the last non-missing value before the start of treatment. Change from Baseline in FBG was calculated as the post-Baseline value minus the Baseline value. The LOCF method was used to impute missing data, in which the last non-missing post-Baseline on-treatment measurement was used to impute the missing measurement. If a participant had missing observation(s) immediately after Baseline, the Baseline observation was not carried forward and was left as missing. Participants were analyzed in a particular treatment week if they had received at least one dose in that treatment week. Based on ANCOVA: Change = treatment + Baseline FPG + renal impairment + prior myocardial infarction history + age category + region.
Time Frame: Baseline; Week 26
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Millimoles per liter (mmol/L)
Arm/Group | Albiglutide 30 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 244 | 240
Millimoles per liter (mmol/L) | -1.42 (0.183) | -0.22 (0.184)

5. Secondary Outcome: Mean Change From Baseline in FPG at Weeks 4, 8, 12, 16, 20, and 26: LOCF
Description: The FPG test measures blood sugar levels after the participant has not eaten (fasted) for 12 to 14 hours. The Baseline FPG value is the last non-missing value before the start of treatment. Change from Baseline in FBG was calculated as the post-Baseline value minus the Baseline value. The LOCF method was used to impute missing data, in which the last non-missing post-Baseline on-treatment measurement was used to impute the missing measurement. If a participant had missing observation(s) immediately after Baseline, the Baseline observation was not carried forward and was left as missing. Participants were analyzed in a particular treatment week if they had received at least one dose in that treatment week.
Time Frame: Baseline; Weeks 4, 8, 12, 16, 20, and 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Albiglutide 30 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 246 | 240
Millimoles per liter (mmol/L)
  Week 4, n=244, 240 | -1.47 (3.054) | -0.84 (2.670)
  Week 8, n=244, 240 | -1.19 (3.115) | -0.82 (3.169)
  Week 12, n=244, 240 | -1.35 (2.930) | -0.81 (3.214)
  Week 16, n=244, 240 | -1.34 (3.070) | -0.49 (3.440)
  Week 20, n=244, 240 | -1.37 (3.198) | -0.62 (3.257)

6. Secondary Outcome: Mean Change From Baseline in Fasting Plasma Glucose (FPG) at Weeks 1, 2, 3, 4, 8, 12, 16, 20, 26, 36, 48, and Week 52: OC
Description: The FPG test measures blood sugar levels after the participant has not eaten (fasted) for 12 to 14 hours. The Baseline FPG value is defined as the last non-missing value prior to treatment. Change from Baseline in FBG was calculated as the post-Baseline value minus the Baseline value. The OC method (no imputation of missing data) was used. If a participant had missing observation(s) immediately after Baseline, the Baseline observation was not carried forward and was left as missing. Participants were analyzed in a particular treatment week if they had received at least one dose in that treatment week.
Time Frame: Baseline; Weeks 1, 2, 3, 4, 8, 12, 16, 20, 26, 36, 48, Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Albiglutide 30 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 246 | 240
Millimoles per liter (mmol/L)
  Week 1, n=219, 217 | -0.82 (2.572) | -0.93 (2.207)
  Week 2, n=226, 223 | -1.28 (2.569) | -0.66 (2.319)
  Week 3, n=230, 219 | -1.25 (3.168) | -0.88 (2.136)
  Week 4, n=231, 226 | -1.55 (2.859) | -0.76 (2.569)
  Week 8, n=221, 210 | -1.24 (2.896) | -0.74 (2.877)
  Week 12, n=224, 216 | -1.46 (2.623) | -0.88 (2.723)
  Week 16, n=214, 204 | -1.41 (2.796) | -0.55 (3.023)
  Week 20, n=207, 191 | -1.51 (2.859) | -1.00 (2.474)
  Week 26, n=200, 177 | -1.54 (2.507) | -0.58 (2.673)
  Week 36, n=186, 149 | -1.42 (2.788) | -0.92 (2.628)
  Week 48, n=165, 140 | -1.08 (2.720) | -0.58 (2.725)
  Week 52, n=149, 114 | -1.06 (2.850) | -0.96 (2.281)

7. Secondary Outcome: Number of Participants Who Achieved Clinically Meaningful HbA1c Response Levels of <6.5% and <7.0% at Week 26: LOCF
Description: The number of participants who acheieved the HbA1c treatment goal (i.e., the number of participants who achieved HbA1c <7% and <6.5% at Week 26) was assessed. The LOCF method was used to impute missing data, in which the last non-missing post-Baseline on-treatment measurement was used to impute the missing measurement. If a participant had missing observation(s) immediately after Baseline, the Baseline observation was not carried forward and was left as missing.
Time Frame: Week 26
Population: ITT Population. Only those participants available at the indicated time point were assessed.
Measure: Number; unit: Participants
Arm/Group | Albiglutide 30 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 242 | 236
Participants
  HbA1c <6.5% | 37 | 29
  HbA1c <7.0% | 103 | 72

8. Secondary Outcome: Number of Participants Who Achieved a Clinically Meaningful Improvement in the HbA1c Response Level of >=1.0%, >=1.5%, and >=2.0% at Week 26: LOCF
Description: The number of participants who a clinically meaningful improvement from Baseline in the HbA1c response level of >=1.0%, >=1.5%, and >=2.0% at Week 26 were assessed. The LOCF method was used to impute missing data, in which the last non-missing post-Baseline on-treatment measurement was used to impute the missing measurement. If a participant had missing observation(s) immediately after Baseline, the Baseline observation was not carried forward and was left as missing.
Time Frame: Week 26
Population: ITT Population. Only those participants available at the indicated time point were assessed.
Measure: Number; unit: Participants
Arm/Group | Albiglutide 30 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 242 | 236
Participants
  HbA1c >=1.0% | 102 | 77
  HbA1c >=1.5% | 49 | 38
  HbA1c >=2.0% | 26 | 17

9. Secondary Outcome: Number of Participants Who Achieved a Clinically Meaningful HbA1c Response Level of <6.5% and <7.0% at Week 52: OC
Description: The number of participants who acheieved the HbA1c treatment goal (i.e., number of participants who achieved HbA1c <7% and <6.5% at Week 26) was assessed. The OC method (no imputation of missing data) was used. If a participant had missing observation(s) immediately after Baseline, the Baseline observation was not carried forward and was left as missing.
Time Frame: Week 52
Population: ITT Population. Only those participants available at the indicated time point were assessed.
Measure: Number; unit: Participants
Arm/Group | Albiglutide 30 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 157 | 118
Participants
  HbA1c <6.5% | 44 | 27
  HbA1c <7.0% | 98 | 61

10. Secondary Outcome: Number of Participants Who Achieved a Clinically Meaningful Improvement in the HbA1c Response Level of >=1.0%, >=1.5%, and >=2.0% at Week 52: OC
Description: The number of participants who a clinically meaningful improvement from Baseline in the HbA1c response level of >=1.0%, >=1.5%, and >=2.0% at Week 52 assessed. The OC method (no imputation of missing data) was used. If a participant had missing observation(s) immediately after Baseline, the Baseline observation was not carried forward and was left as missing.
Time Frame: Week 52
Population: ITT Population. Only those participants available at the indicated time point were assessed.
Measure: Number; unit: Participants
Arm/Group | Albiglutide 30 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 157 | 118
Participants
  HbA1c >=1.0% | 79 | 65
  HbA1c >=1.5% | 43 | 30
  HbA1c >=2.0% | 20 | 15

11. Secondary Outcome: Number of Participants With the Indicated Time to Hyperglycemic Rescue Through Week 52
Description: Hyperglycemic rescue was defined as meeting one of the following criteria, confirmed by a second sample drawn within 7 days and analyzed by the central laboratory: for the Week 2 to Week 4 visit, a single FPG value >=280 milligrams per deciliter (mg/dL); for the >Week 4 and <Week 12 visits, a single FPG value >=250 mg/dL and previous titration for >=4 weeks; for the >=Week 12 and <Week 26 visits, HbA1c >=8.5% and a <=0.5% reduction from Baseline and previous titration for >=4 weeks; for the >=Week 26 and <Week 48 visits, HbA1c >=8.5% and previous titration for >=4 weeks; for the >=Week 48 and <Week 52 visits, HbA1c >=8.0% and previous titration for >=4 weeks. Time to hyperglycemia rescue is the time between the date of first dose and the date of hyperglycemia rescue plus 1 day, or the time between the date of first dose and the date of last visit during active treatment period plus 1 day for participants not requiring rescue.
Time Frame: Week 2 to Week 52
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Albiglutide 30 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 246 | 240
Participants
  Week 2 | 0 | 2
  Week 4 | 0 | 2
  Week 8 | 1 | 3
  Week 12 | 2 | 5
  Week 16 | 5 | 6
  Week 20 | 9 | 14
  Week 26 | 15 | 29
  Week 36 | 25 | 47
  Week 48 | 33 | 53
  Week 52 | 44 | 68

12. Secondary Outcome: Time to Hyperglycemic Rescue Through Week 52
Description: Hyperglycemic rescue was defined as meeting one of the following criteria, confirmed by a second sample drawn within 7 days and analyzed by the central laboratory: for the Week 2 to Week 4 visit, a single FPG value >=280 milligrams per deciliter (mg/dL); for the >Week 4 and <Week 12 visits, a single FPG value >=250 mg/dL and previous titration for >=4 weeks; for the >=Week 12 and <Week 26 visits, HbA1c >=8.5% and a <=0.5% reduction from Baseline and previous titration for >=4 weeks; for the >=Week 26 and <Week 48 visits, HbA1c >=8.5% and previous titration for >=4 weeks; for the >=Week 48 and <Week 52 visits, HbA1c >=8.0% and previous titration for >=4 weeks. Time to hyperglycemia rescue is the time between the date of first dose and the date of hyperglycemia rescue plus 1 day, or the time between the date of first dose and the date of last visit during active treatment period plus 1 day for participants not requiring rescue. This time is divided by 7 to express the result in weeks.
Time Frame: Week 2 to Week 52
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Albiglutide 30 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 246 | 240
Weeks | NA [NA to NA] — There were too few events of hyperglycemia rescue (<50% of participants with events) to calculate the median and confidence interval. | NA [NA to NA] — There were too few events of hyperglycemia rescue (<50% of participants with events) to calculate the median and confidence interval.

13. Secondary Outcome: Change From Baseline in Body Weight at Week 26: LOCF
Description: Change from Baseline was calculated as the post-Baseline weight minus the Baseline weight. The Baseline weight value is defined as the last non-missing value prior to treatment. This analysis used the LOCF method for missing post-Baseline weight values. Weight values obtained after hyperglycemia rescue werre treated as missing and were replaced with pre-rescue values. Based on ANCOVA: Change = treatment + Baseline weight + renal impairment + prior myocardial infarction history + age category + region.
Time Frame: Baseline; Week 26
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Kilograms
Arm/Group | Albiglutide 30 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 244 | 240
Kilograms | -0.79 (0.192) | -0.19 (0.194)

14. Secondary Outcome: Change From Baseline in Body Weight Through Week 26: LOCF
Description: Change from Baseline was calculated as the post-Baseline weight minus the Baseline weight. The Baseline weight value is defined as the last non-missing value prior to treatment. This analysis used the LOCF method for missing post-Baseline weight values. Weight values obtained after hyperglycemia rescue werre treated as missing and were replaced with pre-rescue values.
Time Frame: Baseline; Week 1, Week 2 , Week 3, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Albiglutide 30 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 246 | 240
Kilograms
  Week 1, n=225, 225 | -0.17 (1.215) | 0.12 (1.237)
  Week 2, n=241, 238 | -0.21 (1.317) | -0.02 (1.423)
  Week 3, n=244, 240 | -0.25 (1.392) | 0.01 (1.530)
  Week 4, n=244, 240 | -0.33 (1.456) | 0.09 (1.806)
  Week 8, n=244, 240 | -0.58 (1.768) | 0.02 (1.952)
  Week 12, n=244, 240 | -0.47 (2.055) | 0.03 (2.254)
  Week 16, n=244, 240 | -0.63 (2.197) | -0.08 (2.564)
  Week 20, n=244, 240 | -0.69 (2.556) | -0.07 (2.878)

15. Secondary Outcome: Change From Baseline in Body Weight Through Week 52: OC
Description: Change from Baseline was calculated as the post-Baseline weight minus the Baseline weight. The Baseline weight value is defined as the last non-missing value prior to treatment. This analysis used observed weight values excluding those obtained after hyperglycemia rescue; no missing data imputation was performed.
Time Frame: Baseline; Week 1, Week 2 , Week 3, Week 4, Week 8, Week 12, Week 16, Week 20, Week 26, Week 36, Week 48, and Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Albiglutide 30 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 246 | 240
Kilograms
  Week 1, n=225, 225 | -0.17 (1.215) | 0.12 (1.237)
  Week 2, n=232, 227 | -0.21 (1.339) | -0.01 (1.438)
  Week 3, n=236, 224 | -0.24 (1.404) | 0.03 (1.544)
  Week 4, n=235, 230 | -0.31 (1.466) | 0.10 (1.827)
  Week 8, n=226, 214 | -0.61 (1.800) | 0.05 (2.012)
  Week 12, n=228, 219 | -0.45 (2.091) | 0.16 (2.193)
  Week 16, n=223, 210 | -0.68 (2.226) | 0.07 (2.589)
  Week 20, n=211, 198 | -0.76 (2.619) | 0.09 (2.976)
  Week 26, n=202, 178 | -0.87 (2.856) | -0.04 (3.465)
  Week 36, n=190, 155 | -0.92 (3.551) | 0.01 (2.975)
  Week 48, n=172, 140 | -0.93 (3.829) | 0.07 (3.349)
  Week 52, n=157, 119 | -0.82 (3.931) | 0.31 (3.685)

16. Secondary Outcome: Plasma Concentrations (Conc.) of Albiglutide at Week 8 and Week 16
Description: Sparse population pharmacokinetic (PK) data were collected for population PK and PK/pharmacodynamic (PD) analyses. Participants (par.) who received albiglutide were initiated on a 30 mg weekly dosing regimen. Beginning at Week 4, uptitration of albiglutide was allowed based on glycemic parameters. As such, albiglutide plasma conc. achieved at each sampling time represent a mixed population of par. who received either 30 mg or 50 mg weekly for various durations. The PK and PK/PD of albiglutide were characterized using a population modeling approach. Mean albiglutide plasma conc. observed at Weeks 8 and 16 are presented. Par. came to the clinic at Weeks 8 and 16 without taking albiglutide/matching placebo. The pre-dose PK sample was taken immediately prior to dosing. The Week 8 post-dose sample was taken between Weeks 8 and 10, >=2 days after a dose of medication. The Week 16 post-dose PK sample was taken any time between Weeks 16 and 20, >=2 days after the previous dose of albiglutide.
Time Frame: Week 8 Pre-dose (immediately prior to dose), Week 8 Post-dose (at least 2 days after a dose of medication), Week 16 Pre-dose (immediately prior to dose), and Week 16 Post-dose (at least 2 days after previous dose of albiglutide)
Population: ITT population. Only participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Albiglutide 30 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 228 | 0
nanograms per milliliter (ng/mL)
  Week 8, Pre-dose, n=223 | 3005.80 (1788.544) |
  Week 8, Post-dose, n=220 | 3452.62 (1912.329) |
  Week 16, Pre-dose, n=215 | 2994.15 (1759.161) |
  Week 16, Post-dose, n=205 | 3583.06 (2239.026) |

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the time of study participation consent through Week 60, or the final follow-up visit for participants who discontinued active participation in the study (up to Study Week 60).
Description: On-therapy SAEs and non-serious AEs (events with a start date on or after the first day of study medication [SM] and within 56 days after the end of SM) were collected in members of the Safety Population, comprised of all randomly assigned study participants who received at least one dose of SM.
Arm/Group | Albiglutide 30 mg | Sitagliptin 100 mg
Serious Adverse Events (participants affected / at risk) | 30/249 | 33/246
Other Adverse Events (participants affected / at risk) | 174/249 | 162/246
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Albiglutide 30 mg (N=249) | Sitagliptin 100 mg (N=246)
Atrial fibrillation (Cardiac disorders) | 4 | 1
Coronary artery disease (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 3
Pneumonia (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1
Infected skin ulcer (Infections and infestations) | 0 | 1
Pneumonia necrotising (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1
Pyelonephritis chronic (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectosigmoid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 3
Cerebrovascular disorder (Nervous system disorders) | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Viith nerve paralysis (Nervous system disorders) | 0 | 1
Chest discomfort (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 2
Retinal detachment (Eye disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal ligament ossification (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Chronic obstructive pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis necrotising (Gastrointestinal disorders) | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 1
Arterial thrombosis limb (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Goitre (Endocrine disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Albiglutide 30 mg (N=249) | Sitagliptin 100 mg (N=246)
Urinary tract infection (Infections and infestations) | 21 | 20
Upper respiratory tract infection (Infections and infestations) | 14 | 23
Nasopharyngitis (Infections and infestations) | 14 | 20
Bronchitis (Infections and infestations) | 9 | 7
Influenza (Infections and infestations) | 8 | 7
Gastroenteritis (Infections and infestations) | 5 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 60 | 39
Gout (Metabolism and nutrition disorders) | 11 | 7
Hyperuricaemia (Metabolism and nutrition disorders) | 8 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 7 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 25 | 16
Constipation (Gastrointestinal disorders) | 15 | 6
Nausea (Gastrointestinal disorders) | 12 | 8
Haemorrhoids (Gastrointestinal disorders) | 6 | 3
Dyspepsia (Gastrointestinal disorders) | 5 | 9
Gastritis (Gastrointestinal disorders) | 5 | 7
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 10
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 6
Oedema peripheral (General disorders) | 13 | 8
Injection site reaction (General disorders) | 10 | 1
Fatigue (General disorders) | 5 | 2
Injection site pruritus (General disorders) | 5 | 0
Injection site haematoma (General disorders) | 3 | 6
Hypertension (Vascular disorders) | 14 | 19
Hypotension (Vascular disorders) | 3 | 5
Renal failure (Renal and urinary disorders) | 12 | 10
Renal impairment (Renal and urinary disorders) | 6 | 8
Headache (Nervous system disorders) | 8 | 11
Dizziness (Nervous system disorders) | 8 | 5
Diabetic retinopathy (Eye disorders) | 12 | 9
Cataract (Eye disorders) | 9 | 5
Anaemia (Blood and lymphatic system disorders) | 16 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Vertigo (Ear and labyrinth disorders) | 3 | 5
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.